CLINICAL TRIAL: NCT06977997
Title: Temporomandibular Disorders: Knowledge, Attitude, and Practice Among Dentists in Egypt: A Cross-sectional Study
Brief Title: Temporomandibular Disorders Knowledge, Attitude, and Practice in Egypt
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Emad Ibrahim, Post-graduate student, Cairo University
Other Study IDs: TMD Knowledge
Record Dates: First submitted 2025-05-03; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: KAP survey — 33 questions to assess knowledge, attitude, and practice of dentists in Egypt regarding TMD

SUMMARY:
Primary objective:

Evaluate the level of knowledge, and attitude of dental practitioners in Egypt.

Secondary objectives:

1. Evaluate the need for continuing dental education in the field of TMD.
2. Describe referral process practiced by dental practitioners.
3. Describe the procedures practiced by the dental practitioners for diagnosis and management of TMD.

DETAILED DESCRIPTION:
To the best of our knowledge, no studies have been conducted to evaluate the knowledge, attitudes, and practices of Egyptian dental practitioners regarding TMD. Knowledge can be categorized into essential sections for assessment, including aetiology, diagnosis, and management. Etiology and diagnosis are fundamental for providing effective management, which in turn reflects the quality of care received by patients. Evaluating the KAP of the GDPs regarding TMD can be applied to assess areas of knowledge shortfall and correlation between levels of knowledge and attitudes with years of practice experience and specialty. This can also reflect how effective the training at the dental school, as well as the postgraduate training, has been in this context. Besides, practice illustrates how practitioners apply their knowledge and attitudes to make appropriate patient diagnoses and management, as well as to describe the referral process

ELIGIBILITY:
Inclusion Criteria:

1. Gender: both males and females.
2. Dentists practicing the profession in Egypt
3. General practitioners or specialists

Exclusion Criteria:

1-Undergraduate students

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dental practitioners practicing the profession in Egypt
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
level of knowledge, and attitude of dental practitioners in Egypt. | Immediately after the dentists complete the questionnaire
  knowledge, attitude will be assessed using questionnaire consisted of four domains: demographics, knowledge, attitude, and practice. content validity and reliability will be performed. Continuous data was explored for normality using Kolmogrov Smirnov test and Shapiro Wilk test.Continuous data showed non-parametric distribution and was described using mean, standard deviation, median and range. knowledge score range from 1 to 14, and attitude score range from 0 to 5. where higher scores indicate a higher knowledge and attitude levels

SECONDARY OUTCOMES:
The percentage of each speciality to whom the dentists participating to the questionnaire are referring TMD patients using their answers to the questionnaire | Immediately after the dentists complete the questionnaire
  descriptive analysis using categorical and binary data will be presented as frequency and percentage
percentage of different treatment modalities offered by participant to TMD patient assessed by their answers to the questionnaire | Immediately after the dentists complete the questionnaire
  descriptive analysis using categorical and binary data will be presented as frequency and percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aldrigue RH, Sanchez-Ayala A, Urban VM, Pavarina AC, Jorge JH, Campanha NH. A Survey of the Management of Patients with Temporomandibular Disorders by General Dental Practitioners in Southern Brazil. J Prosthodont. 2016 Jan;25(1):33-8. doi: 10.1111/jopr.12255. Epub 2015 Jan 5. PMID 25557469
- [Background] Al-Huraishi HA, Meisha DE, Algheriri WA, Alasmari WF, Alsuhaim AS, Al-Khotani AA. Newly graduated dentists' knowledge of temporomandibular disorders compared to specialists in Saudi Arabia. BMC Oral Health. 2020 Oct 7;20(1):272. doi: 10.1186/s12903-020-01259-4. PMID 33028397
- [Background] Celakil T, Saruhanoglu A. Knowledge and Attitude Toward Temporomandibular Disorders: A Survey in Istanbul. Turk J Orthod. 2022 Mar;35(1):39-45. doi: 10.5152/TurkJOrthod.2022.21170. PMID 35370133